CLINICAL TRIAL: NCT05710237
Title: Does Psilocybin Require Psychedelic Effects to Treat Depression? A 4-Week, Double-Blind, Proof-of-Concept Randomized Controlled Trial
Brief Title: Does Psilocybin Require Psychedelic Effects to Treat Depression?
Acronym: PSI-RIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 080-2022
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Treatment-resistant Depression
Keywords: Psilocybin; Psychedelics; Treatment-resistant depression; Clinical trial
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Psilocybin; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, their families, the study investigator, study therapists, and research assistants carrying out assessments will be concealed from allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Risperidone 1 mg plus Psilocybin 25 mg (Experimental): Risperidone 1 mg plus Psilocybin 25 mg
  Interventions: Drug: Psilocybin 25 mg; Drug: Risperidone 1 MG
- Placebo plus Psilocybin 25 mg (Experimental): Placebo plus Psilocybin 25 mg
  Interventions: Drug: Psilocybin 25 mg; Drug: Placebo
- Risperidone 1 mg plus Placebo (Active Comparator): Risperidone 1 mg plus Placebo
  Interventions: Drug: Risperidone 1 MG; Drug: Placebo

INTERVENTIONS:
Drug: Psilocybin 25 mg — The psilocybin used in this study meets quality specifications suitable for human research use. The active drug is encapsulated using a hydroxypropyl methylcellulose (HPMC) capsule and contains 25 mg of psilocybin. The psilocybin will be administered once during the trial in combination with either risperidone 1 mg or place. It will also be administered in conjunction with supportive therapy.
  Arms: Placebo plus Psilocybin 25 mg; Risperidone 1 mg plus Psilocybin 25 mg
Drug: Risperidone 1 MG — The risperidone is encapsulated using a cellulose capsule and contains 1 mg of risperidone. The risperidone will be administered once during the trial in combination with either psilocybin 25 mg or placebo. It will also be administered with supportive therapy.
  Arms: Risperidone 1 mg plus Placebo; Risperidone 1 mg plus Psilocybin 25 mg
Drug: Placebo — The placebo will be administered once during the trial in combination with either risperidone 1 mg or psilocybin 25 mg.
  Arms: Placebo plus Psilocybin 25 mg; Risperidone 1 mg plus Placebo

SUMMARY:
Psilocybin, the chemical component of "magic mushrooms", has been administered with psychotherapy in several randomized clinical trials (RCTs) showing large and sustained antidepressant effects. In healthy volunteers, the psychedelic effects of psilocybin have been shown to be blocked by administration of serotonin (5HT)2A receptor antagonists such as risperidone.

The purpose of this "double dummy" proof-of-concept trial is to evaluate whether psilocybin's antidepressant effects are dependent on its psychedelic effects. Sixty participants with treatment-resistant depression will be randomly assigned to one of three groups: 1) Psilocybin 25 mg plus risperidone 1 mg; 2) Psilocybin 25 mg plus placebo; and 3) Placebo plus risperidone 1 mg. The investigator's hypothesize that the combination of psilocybin and risperidone will be well tolerated, safe, and will block the psychedelic effects of psilocybin in patients diagnosed with treatment-resistant depression.

DETAILED DESCRIPTION:
This study is a three-arm, 4-week, double blind, proof-of concept RCT for investigating psilocybin-assisted psychotherapy (PAP) administered with risperidone in treating TRD. This three-arm "double dummy" design allows for an assessment of risperidone's anti-psychedelic effects, while allowing for an assessment of psilocybin's antidepressant effects alone and combined with risperidone, compared to an "active placebo" (i.e. placebo plus risperidone 1 mg).

Overview of Study Design:

A study team member will obtain informed consent from interested participants prior to study activities being initiated. Following this, participants will undergo a screening assessment where they will complete lab tests, and clinical and psychiatric assessments to determine eligibility. Following the screening visit, eligible participants will undergo a washout period where they will be tapered off concomitant medication over a period of 4 to 6 weeks. The length of the tapering period will depend on the type of medication the participant is being tapered off (based on the half-life of the medication) and the participant's preference for the length of the tapering period. Most medications will require a minimum of a 2-week tapering period before the baseline, with the exception of fluoxetine, which will require a minimum of 4-weeks. Additional time may be added at the discretion of the study investigator. During the tapering period, the study psychiatrist will see participants weekly (V1a, V1b, etc.) for at least 4 weeks to monitor for withdrawal and worsening of depressive symptoms and suicidality. Suicidality will be closely monitored using the Columbia Suicide Severity Rating Scale (C-SSRS). Participants and their family members/carers will be educated on the signs and symptoms of worsening depression and suicidality and will be given contact details of the study team in case of major decline in mental state.

At the Baseline visit (V2), which occurs the day before the dosing session, participants will complete clinical measures, and undergo a preparatory session (up to 4 hours) with the study therapists. These sessions will build a therapeutic alliance, provide psychoeducation about, and set intentions for, the psilocybin session. To reduce participant burden, baseline can be broken up into multiple days, however all assessments must be completed within 7-days of the intervention. Ideally, baseline occurs the day before the intervention is administered.

The psilocybin session (Day 0 [V3]) will last 5 to 6 hours and will be conducted in the existing psychedelic treatment suite developed at the Centre for Addiction and Mental Health (CAMH) Mood Disorder Service by Dr. Husain (PI). Two trained study therapists will be supporting each participant during the dosing session. Participants will receive psilocybin 25 mg plus risperidone 1 mg, or psilocybin 25 mg plus placebo, or placebo plus risperidone 1 mg. All participants will receive 10 hours of manualized supportive psychotherapy (which includes the 5-6 hour dosing session). After 5 hours of dose administration, participants will be evaluated for safety by the study psychiatrist and discharged home in the company of a caregiver or a family member.

After the dosing session, participants will be seen for two 1-hour integration sessions (Day 1 [V4], Week 1 [V5]). Thereafter, participants will be followed-up after 2 [V6], 3 [V7] and 4 weeks [V8] post-dosing (see Figure 1). A study psychiatrist will be available throughout the duration of the RCT to respond to any concerns or changes in mental/physical state. Participants will not start other interventions for MDD during the study.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient adults 18 to 65 years old;
* Able to provide informed consent and read and communicate in English;
* Primary DSM-5 diagnosis of non-psychotic MDD, single or recurrent, based on the Structured Clinical Interview for DSM-5 (SCID-5);
* Diagnosis of treatment-resistant depression defined as a baseline HamD-17 score > 14 and have not responded to two or more separate trials of antidepressants at an adequate dosage and duration (an antidepressant resistance rating score of three or more is considered an adequate trial) based on the Antidepressant Treatment History Form (ATHF); there is no upper limit on the number of treatment failures;
* Ability to take oral medication;
* All bloodwork within normal limits or assessed as not clinically significant by study physicians and an eGFR above 40mL/min/1.73m2;
* Individuals who are capable of becoming pregnant: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation;
* Willing to and have tapered off current antidepressant and antipsychotic medications for a minimum of 2-weeks (or more depending on the medication) prior to baseline and for the duration of the study and whose physician confirms that it is safe for them to do so; AND
* Willing to and have tapered off current inhibitors of 5'-diphospho-glucuronosyltransferase (UGT)1A9 and 1A10, aldehyde dehydrogenase inhibitors (ALDHs) and alcohol dehydrogenase inhibitors (ADHs) for a minimum of 2-weeks (or more depending on the medication) prior to baseline and for the duration of the study and whose physician confirms that it is safe for them to do so;

Exclusion Criteria:

* Pregnant or individual's that intend to become pregnant during the study or are breastfeeding;
* Treatment with another investigational drug or other intervention within 30 days of screening;
* Have initiated psychotherapy in the preceding 12 weeks prior to screening;
* Have a DSM-5 diagnosis of substance use disorder (recreational use of tobacco, alcohol, cannabis and prescribed opioids are permitted) within the preceding 6-months;
* Have active suicidal ideation with intent and plan as determined by item 3 of the HamD-17;
* Any DSM-5 lifetime diagnosis of a schizophrenia-spectrum disorder, obsessive-compulsive disorder, psychotic disorder (unless substance induced or due to a medical condition), bipolar I or II disorder, paranoid personality disorder, borderline personality disorder, or neurocognitive disorder as determined by medical history and the SCID-5 clinical interview;
* Any first-degree relative with a diagnosis of schizophrenia-spectrum disorder; psychotic disorder (unless substance-induced or due to a medical condition); or bipolar I or II disorder;
* Presence of a relative or absolute contraindication to psilocybin, including a drug allergy, recent stroke history, uncontrolled hypertension, low or labile blood pressure, recent myocardial infarction, cardiac arrhythmic, severe coronary artery disease, or moderate to severe renal or hepatic impairment;
* Presence of baseline prolonged QTc or Torsade de Pointes as measured by the ECG or a history of long QTc syndrome or related risk factors;
* History of allergy or contraindication to risperidone including insulin-dependent diabetes, history of hypoglycemia on oral hypoglycemic agent(s)
* Lifetime use of serotonergic psychedelic drugs; OR
* Any other clinically significant physical illness including chronic infectious diseases or any other major concurrent illness that, in the opinion of the investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if they take part in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility of administering psilocybin (25mg) with risperidone (1mg) | 4 weeks
  Percentage of participants recruited, randomized, and retained.
Tolerability and safety of administering psilocybin (25mg) with risperidone (1mg) | 4 weeks
  Frequency of dropouts attributed to adverse effects or serious adverse events

SECONDARY OUTCOMES:
Subjective psychedelic effects as measured by the 5-Dimensional Altered States of Consciousness (5D-ASC) Rating Scale | Visit 3 (Day 0)
  A visual analogue scale (0-100 millimeters in length) with higher scores indicating more intense effects.

OTHER OUTCOMES:
Change in the Montgomery-Åsberg Depression Rating Scale (MADRS) from Baseline to 1-week post-treatment. | Baseline (Day -1) to visit 5 (Day 7)
  The Montgomery-Åsberg Depression Rating Scale is a clinician-rated scale that measures depression severity. It is 10-items which are scored from 0 (not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60.
  Higher scores represent a more severe condition.

CONTACTS AND LOCATIONS:
Overall Officials: M. Ishrat Husain, MBBS, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT05710237/Prot_SAP_002.pdf